CLINICAL TRIAL: NCT04912648
Title: FEmale Metabolic Risk and Androgens: an Irish Longitudinal (FEMAIL) Study
Acronym: FEMAIL
Status: Recruiting | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 20/49
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Hyperandrogenism; Metabolic Disease; Sex Hormones Adverse Reaction
MeSH Terms: conditions — Hyperandrogenism; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum; urine; saliva; muscle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women age 18 years and older: * baseline anthropometry
  * bloods for metabolic phenotype; targeted and nontargeted Metabolomics
  * saliva and urine for steroid Metabolomics
  * bioimpedance
  * muscle biopsy for transcriptomics
  Interventions: Other: Longitudinal follow up

INTERVENTIONS:
Other: Longitudinal follow up — Repeat follow up at 3,5 and 10 years

SUMMARY:
Androgen excess is the cardinal biochemical feature of polycystic ovary syndrome (PCOS), a lifelong metabolic disorder affecting 10% of women. Serum testosterone correlates with insulin resistance in women, however, there is an urgent need to improve our understanding of the association between androgens and the risk of type 2 diabetes. Recently, a new subclass of androgenic steroids known as 11-oxygenated androgens has been identified. Utilising highly sensitive liquid chromatography-tandem mass spectrometry (LC-MS/MS) techniques, our group has recently demonstrated that 11-oxygenated steroids are the predominant androgens in both health controls and women with PCOS, and that these correlate closely with markers of insulin resistance. The bioactive 11-oxygenated androgen 11-ketotestosterone (11KT) binds and activates the androgen receptor with equal affinity to testosterone, yet nothing is known about its impact on metabolism or glucose homeostasis. Intriguingly, unlike testosterone, 11-oxygenated androgens do not decline with age in women, and, therefore, may mediate an increased risk of T2DM in women across their life course. Therefore, this previously ignored androgen class is likely of major importance in female metabolic health, and may represent a novel metabolic risk factor and biomarker. However, 11-oxygenated androgens are not currently measured in routine clinical practice. To date, no population-based or human in vivo physiology studies have examined the association between 11-oxygenated androgens, glucose metabolism and diabetes risk in women, despite the high prevalence of PCOS in the female population. There is emerging evidence, even in women without a confirmed history of PCOS, that the levels of androgens over time correlate with their likelihood of developing metabolic and cardiovascular disease. This has not been studied to date in a prospective manner in healthy women in the background population using long term follow up data.

DETAILED DESCRIPTION:
Clinical questionnaire and baseline anthropometry:

Study investigators will complete a standardised case record form, with information obtained on relevant medical history, medications and anthropometric assessment (height, weight, body mass index, blood pressure, weight circumference). Body composition will be assessed using a portable bioimpedance machine (Tanita MC-780MA-S Portable). We will also obtain information on education level and household income. Participants will complete a standardised QOL questionnaire.

Serum, urine and saliva sampling:

Fasting bloods will be drawn for assessment of metabolic phenotype including glucose, insulin, lipid profile, full blood count, renal and liver biochemistry and HbA1C. Serum samples will also be obtained for measured of the steroid and non-targeted metabolome. Urine and saliva samples will be obtained for assessment of steroid metabolomics.

Targeted steroid metabolome profiling:

Serum, urinary and salivary multi-steroid profiling including classic and 11-oxygenated androgens will be performed using highly sensitive liquid chromatography tandem mass spectrometry (LC-MS/MS). Furthermore, we will analyse the 24-h urine steroid metabolome, allowing for determination of 24-h net androgen output from classic and 11-oxygenated pathways (26). Analysis will be carried out by LC-MS/MS multi-steroid profiling. Multi-steroid profiling approaches have been developed and optimised at the University of Birmingham Steroid Metabolome Analysis Core (SMAC), where samples will be measured under the supervision of Professor Wiebke Arlt.

Non-targeted serum metabolomics:

The global non-targeted serum metabolome will be profiled at the Phenome Centre Birmingham under the supervision of Professor Warwick Dunn (co-applicant). Samples will be analysed applying Ultra Performance Liquid Chromatography (Ultimate3000RS; Thermo Scientific, Hemel Hempstead, UK) interfaced to an electrospray mass spectrometry (Q Exactive, Thermo Scientific, Hemel Hempstead, UK).

Muscle biopsy:

Under local anaesthetic and without using scalpel incision, muscle biopsies will be obtained from the vastus lateralis muscle of the leg in each participant. These will be performed using a Bard biopsy needle gun, with suction applied to increase tissue yield.

Recruitment:

Patients will be recruited via local advertising in Beaumont Hospital and RCSI Medical School.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Ability to provide informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding at the time of planned recruitment
* History of significant renal (eGFR<30) or hepatic impairment (AST or ALT >two-fold above ULN; pre-existing bilirubinaemia >1.2 ULN)
* The investigators will retain the right not to recruit potential participants with severe health disorders which may impact on their ability to participate in the study; these may include, but are not limited to, metastatic cancer, severe cardio-respiratory disease or other life-limiting health disorders
* Participants who have participated in another research study involving an investigational medicinal product in the 12 weeks preceding the planned recruitment
* Glucocorticoid use via any route within the last six months
* Current intake of drugs known to impact upon steroid or metabolic function or intake of such drugs during the six months preceding the planned recruitment
* Use of combined oral hormonal contraception in the three months preceding the planned recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female 46XX
Study Population: Women meeting the above inclusion criteria without exclusion criteria
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of sex hormone profiles and the metabolome of women across the lifespan with risk of metabolic dysfunction, cardiovascular disease and quality of life. | 3 years

SECONDARY OUTCOMES:
Development of risk prediction models for development of diabetes in women | 5 years
Establishment of the longitudinal FEMAIL study database | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Royal College of Surgeons in Ireland, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be made available after consideration of individual access requests, in line with data protection laws and participant consent